CLINICAL TRIAL: NCT03044210
Title: Metabolic Study of Cockayne Syndrome
Acronym: METABO-CS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pas assez de patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6372
Record Dates: First submitted 2017-01-16; First posted 2017-02-06 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Cockayne Syndrome
Keywords: Rest energetic cost measured by indirect calorimetry; Hormonal axis; Mitochondrial oxidative phosphorylation; Basal metabolism
MeSH Terms: conditions — Cockayne Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cockayne patients (Other): Interventions performed:
  * blood sample
  * urinary collection
  * metabolic evaluation
  * clinical evaluation
  Interventions: Other: Metabolic evaluation
- Control subjects (Other): Interventions performed:
  * urinary collection
  * metabolic evaluation
  * clinical evaluation
  Interventions: Other: Metabolic evaluation

INTERVENTIONS:
Other: Metabolic evaluation — * diet assessment
  * biological evaluation
  * clinical evaluation
  * metabolic evaluation (calorimetry)

SUMMARY:
Cockayne syndrome (CS) is related to defective DNA transcription and/or repair and belongs to the family of Nucleotide Excision Repair. It is an autosomal recessive multisystemic disorder characterized by mental retardation, microcephaly, severe growth failure with lipoatrophia, sensorial impairment, cutaneous photosensitivity, dental decay, enophtalmios. The disease is progressive causing severe impairments but there's currently no therapeutics for the disease.

Growth failure, feeding difficulties and lipoatrophia are prognostic keys of CS but physiopathology is unknown.

According to preliminary assays, our goal is to test the hypothesis that cachexia is due to hypometabolism. We also want to test the potential link between this basal metabolism modification and mitochondrial dysfunction and somatotrope axis, and correlation between the basal metabolism degree and global severity of the disease.

ELIGIBILITY:
Cockayne patients:

Inclusion criteria :

* Male and female with cockayne syndrome
* Age>6 months

Exclusion criteria:

* Intercurrent diseases
* Subject in period of exclusion
* Pregnancy and breastfeeding

Control subjects :

Inclusion criteria :

* Sister or brother of Cockayne patients
* Age>6 months

Exclusion criteria:

* Intercurrent diseases
* Subject in periods of exclusion
* Pregnancy and breastfeeding

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Rest energetic cost measured by indirect calorimetry compared to calculated Black equation | Day 0

SECONDARY OUTCOMES:
Rest energetic cost measured by indirect calorimetry compared to calculated theorical equations | Day 0
Hormonal axis evaluation and mitochondrial activity measured by level of hormones and lactates/pyruvates in blood | Day 0
Respiratory quotient measured by indirect calorimetry | Day 0
Fat mass and lean mass measured by impedancemetry | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude SPITZ, MD, Principal Investigator — Hôpitauc Universitaires de Strasbourg
Locations (1):
- Centre d'Investigation Clinique, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No